CLINICAL TRIAL: NCT02146118
Title: A Phase II Study to Assess Efficacy of Combined Treatment With Erlotinib (Tarceva) and Silybin-phytosome (Siliphos) in Patients With EGFR(Epidermal Growth Factor Receptor) Mutant Lung Adenocarcinoma
Brief Title: A Phase II Study to Assess Efficacy of Combined Treatment With Erlotinib (Tarceva) and Silybin-phytosome (Siliphos) in Patients With EGFR Mutant Lung Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MedicalLogic (Industry)
Collaborators: Kosin University Gospel Hospital (Other)
Responsible Party: Principal Investigator, Chang-gyu Choi, Manager, MedicalLogic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLB-001
Record Dates: First submitted 2014-05-07; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Erlotinib; Silybin-phytosome; EGFR mutant lung adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; silybin-phytosome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib and Silibin (Experimental)
  Interventions: Drug: Erlotinib; Dietary Supplement: Silybin-phytosome

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg/day q 4 weeks
  Other Names: Tarceva
Dietary Supplement: Silybin-phytosome — Silybin-phytosome 1g bid/day q 4 weeks
  Other Names: Siliphos

SUMMARY:
1. Title and stage of study A Phase II Study to Assess Efficacy of Combined Treatment with Erlotinib (Tarceva) and Silybin-phytosome (Siliphos) in Patients with EGFR mutant lung adenocarcinoma
2. Endpoints Primary Endpoint : tumour response rate Secondary Endpoint : progression-free survival, overall survival, and safety assessment
3. Study Rationale Even though it is commonly accepted that EGFR TKIs are effective to EGFR mutation positive lung cancer patients, still remains its resistance issue.

   The Silybin which is extract from mugwort bean Thistle and used for hepatoprotective drug for a long time with very low adverse events in Eastern countries. Recently, there are some reports regarding its anti-cancer effects through several preclinical studies.

   The safety of Siliphos which is developed agent from silybin for improving intestinal absorption was demonstrated in PhaseⅠtrial.

   Recently investigators found out Silybin is effective for blocking EGFR signal in different mechanism from Erlotinib and it can be expected additional impact with combination therapy with preclinical data.

   Our research team can expect to improve Lung cancer treatment if the combination therapy (Silybin_Erlotinib) improves patients' response and Overall survivor.
4. Treatment method Erlotinib (Tarceva 150 mg/day) and Silybin (Siliphos 1g bid/day) q 4 weeks
5. Assessment criteria For toxicity assessment, posttreatment recurrence and survival rates will be investigated based on NCI-CTCAE ver 4.0 and RTOG. Efficacy assessment will be conducted through measurement of lesions by CT and RECIST criteria. Overall survival (OS), progression-free survival (PFS), and time to tumour progression (TTP) will be estimated using a Kaplan-Meier analysis. In addition, effect of pre-treatment T790M on response and PFS will be analyzed.

DETAILED DESCRIPTION:
1. Title and stage of study

   A Phase II Study to Assess Efficacy of Combined Treatment with Erlotinib (Tarceva) and Silybin-phytosome (Siliphos) in Patients with EGFR mutant lung adenocarcinoma
2. Endpoints

   Primary Endpoint : tumour response rate Secondary Endpoint : progression-free survival, overall survival, and safety assessment
3. Inclusion/exclusion criteria

   Inclusion criteria
   1. Histological or cytologic diagnosis of stage IV lung adenocarcinoma and confirmed EGFR mutation
   2. Patients who have not received chemotherapy before. However, patients who received postoperative adjuvant chemotherapy more than 6 months ago are eligible.
   3. Patients with a lesion that can be measured a response-evaluation according to the RECIST criteria (at least one evaluable lesion)
   4. Patients aged 20 years or older
   5. ECOG performance status score of 0, 1 or 2
   6. Expected lifetime of ≥3 months
   7. Adequate bone marrow and liver functions maintained

      1. Neutrophil count: > 1,500/㎕
      2. Platelet count: > 100,000/㎕
      3. Hb: > 9.0g/dL
      4. AST/ALT: < 2.0 x upper normal limit
      5. Bilirubin: < 1.25 x upper normal limit
   8. Patients or their legally acceptable representatives must complete a written consent before initiation of the study and patients can comply with requirements for the study

   Exclusion criteria
   1. Symptomatic central nervous system (CNS) malignant tumor or metastasis. However, the patients who are treated for CNS metastasis can be enrolled if their disease is radiologically stable and asymptomatic. Asymptomatic patients without a history of CNS metastasis do not need screening.
   2. Evidence of severe or uncontrolled systemic diseases at the investigator's discretion (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal diseases)
   3. Patients who have been treated with EGFR inhibitors before
   4. Patients treated with other investigational products or unapproved drugs within 28 days before enrollment in this study
   5. Pregnant and lactating women, and patients of childbearing who do not agree to use contraception
   6. Patients ineligible for the study at the investigator's discretion
4. Study Rationale

   Even though it is commonly accepted that EGFR TKIs are effective to EGFR mutation positive lung cancer patients, still remains its resistance issue.

   The Silybin which is extract from mugwort bean Thistle and used for hepatoprotective drug for a long time with very low adverse events in Eastern countries. Recently, there are some reports regarding its anti-cancer effects through several preclinical studies.

   The safety of Siliphos which is developed agent from silybin for improving intestinal absorption was demonstrated in PhaseⅠtrial.

   Recently investigators found out Silybin is effective for blocking EGFR signal in different mechanism from Erlotinib and it can be expected additional impact with combination therapy with preclinical data.

   Our research team can expect to improve Lung cancer treatment if the combination therapy (Silybin_Erlotinib) improves patients' response and Overall survivor.
5. Treatment method

   Erlotinib (Tarceva 150 mg/day) and Silybin (Siliphos 1g bid/day) q 4 weeks
6. Assessment criteria

   For toxicity assessment, posttreatment recurrence and survival rates will be investigated based on NCI-CTCAE ver 4.0 and RTOG. Efficacy assessment will be conducted through measurement of lesions by CT and RECIST criteria. Overall survival (OS), progression-free survival (PFS), and time to tumour progression (TTP) will be estimated using a Kaplan-Meier analysis. In addition, effect of pre-treatment T790M on response and PFS will be analyzed.
7. Statistical method Object response rate (ORR) will be reported with its 2-sided 95% confidence interval. If the evaluable number of subject is 42 and number of response is 25 or more, this study certainly imply that this treatment has an efficacy worthy of further investigation, perhaps in a Phase III randomized trial.

Progression Free Survival (PFS) is defined as the time from beginning of treatment until object disease progression as defined by RECIST or death. Patient who have not progressed or died at the time of the statistical analysis will be censored at the time of their last evaluable RECIST assessment. Kaplan-Meier plots of PFS and estimated of median PFS will be presented.

Overall survival (OS) is defined as the time from beginning of treatment until death by any cause. Patient who have not died at the time of the data cut-off, or are lost to follow up will be censored at the time they were last known to be alive. Kaplan-Meier plots of OS and estimated of median PFS will be presented.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histological or cytologic diagnosis of stage IV lung adenocarcinoma and confirmed EGFR mutation
* 2. Patients who have not received chemotherapy before. However, patients who received postoperative adjuvant chemotherapy more than 6 months ago are eligible.
* 3. Patients with a lesion that can be measured a response-evaluation according to the RECIST criteria (at least one evaluable lesion)
* 4. Patients aged 20 years or older
* 5. ECOG performance status score of 0, 1 or 2
* 6. Expected lifetime of ≥3 months
* 7. Adequate bone marrow and liver functions maintained

  1. Neutrophil count: > 1,500/㎕
  2. Platelet count: > 100,000/㎕
  3. Hb: > 9.0g/dL
  4. AST/ALT: < 2.0 x upper normal limit
  5. Bilirubin: < 1.25 x upper normal limit
* 8. Patients or their legally acceptable representatives must complete a written consent before initiation of the study and patients can comply with requirements for the study

Exclusion Criteria:

* 1. Symptomatic central nervous system (CNS) malignant tumour or metastasis. However, the patients who are treated for CNS metastasis can be enrolled if their disease is radiologically stable and asymptomatic. Asymptomatic patients without a history of CNS metastasis do not need screening.
* 2. Evidence of severe or uncontrolled systemic diseases at the investigator's discretion (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal diseases)
* 3. Patients who have been treated with EGFR inhibitors before
* 4. Patients treated with other investigational products or unapproved drugs within 28 days before enrollment in this study
* 5. Pregnant and lactating women, and patients of childbearing who do not agree to use contraception
* 6. Patients ineligible for the study at the investigator's discretion

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-09 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Tumour response rate | 12 months
  Efficacy assessment will be conducted through measurement of lesions by CT and RECIST criteria.

SECONDARY OUTCOMES:
Safety assessment | 12 months
  For toxicity assessment, posttreatment recurrence and survival rates will be investigated based on NCI-CTCAE ver 4.0 and RTOG.

CONTACTS AND LOCATIONS:
Overall Officials: Tae won Jang, Dr, Study Director — Kosin University Gospel Hospital
Locations (1):
- Gosin University Gospel Hospital, Busan, Busan, South Korea